CLINICAL TRIAL: NCT06968377
Title: Preliminary Clinical Evaluation of a Novel Airborne Pathogen Containment Device Design: Randomized Open-label Equivalence Trial of Patient Safety and Acceptability During Endotracheal Intubation.
Brief Title: The COVID Dome Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IWK Health Centre (Other)
Responsible Party: Principal Investigator, Dr. Ana Sjaus, Associate Chief - Department of Women's & Obstetric Anesthesia, IWK Health Centre, IWK Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1027983; 1026879 (Other Grant/Funding Number: Department of Anesthesia, Pain Management and Perioperative Medicine, Dalhousie University); 381288 (Registry Identifier: Health Canada - Medical Devices Directorate)
Record Dates: First submitted 2025-05-06; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Medical Device; Medical Device Performance; Aerosol Generating Procedure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dome (Experimental): The device is a large, bubble-like dome made of clear plastic through which doctor and nurse can care for the patient during surgery.
  Interventions: Device: A novel airborne pathogen containment device.
- No dome (No Intervention): Standard care during surgery.

INTERVENTIONS:
Device: A novel airborne pathogen containment device. — The dome is placed over the patient's head during the full duration of a surgery (intubation and extubation included) as a method of preventing infection transmission through airborne aerosols throughout a hospital.
  Arms: Dome

SUMMARY:
The aim of this study is to test a bubble-like dome (made of clear plastic) being placed over patients' heads during surgery as a tool to prevent the spread of germs through the air in hospitals.

The researchers are interested in the following outcomes:

* How the device affects the patients' experience of surgery.
* The impact of the device on how long it takes to place a breathing tube, blood pressure, heart rate and oxygen levels of the patient.

Researchers will compare the outcomes across patients using the device and patients not using the device. This will be done by randomly (by chance) assigning participants undergoing surgery to group 1 (using the bubble-like dome device) or group 2 (not using the device).

Participants will:

* Tell the researchers or your anesthesia doctor about any problems that you experience that you think might be related to participating in the study.
* Fill out a 10-minute survey regarding your experience with the dome after surgery.
* If you did not try the dome before going to sleep, you will be able to watch a video of the dome in use and answer questions based on the video
* Be video recorded with your time with the dome.

DETAILED DESCRIPTION:
Background and Rationale Pandemic spread of COVID-19 presents an unprecedented challenge for health care systems around the world. A highly infectious respiratory virus with long incubation, asymptomatic transmission and environmental stability, SARS-CoV-2 places health care workers (HCWs) at risk of contracting the infection and transmitting it to patients.[1] The early problems with personal protective equipment (PPE) supply have led to a renewed urgency to develop a number of different layers of mitigation. Together, these would offer equitable protection and rational supply management. Central to PPE use are questions related to the type (droplets, aerosol or contact) and magnitude (viral load) of the risk in specific situations. [2][3] Given the unprecedented transmissibility of the newer variants, there is an interest in further mitigating potential exposure. This would be particularly relevant for procedures that limit ability to apply source control such as masking the infectious individual.

Transmission of SARS-CoV-2 is currently understood to occur primarily by respiratory droplets (> 20 microns in diameter), aerosols (< 5 microns) and direct mucosal contact with respiratory secretions.[4] While aerosolization during aerosol generating medical procedures (AGMP) is still a significant focus of infection control protocols, it is increasingly clear that physiologic aerosolization is at least as important. Aerosols containing viral particles can remain suspended and viable in the air for up to 3 hours under experimental conditions.[5] They can be carried by airstream and, when inhaled, be deposited into the lungs as deep as the alveoli. In the setting of perioperative care, AGMPs are administration of oxygen by high-flow nasal cannula, non-invasive positive pressure ventilation, endotracheal intubation and extubation. To minimize aerosol contamination of the facility, Canadian Anesthesiologists' Society and American Society of Anesthesiologists recommend that airway management should ideally be performed in a negative pressure room, while avoiding direct flow of pressurized gas into the patient's airway.[6-8] This is achieved by limiting flow rate during preoxygenation, ensuring deep muscle relaxation to avoid cough, applying a HEPA filter to the endotracheal tube and inflating the tracheal cuff prior to connecting the ventilator circuit. Very few operating rooms in Canada (and worldwide) are built as isolation rooms. Furthermore, the risk to HCWs who are in the immediate vicinity of the source, performing the procedure, is however, minimally mitigated by these measures.

The ability to apply source control and contain the spread of aerosol at the time of AGMP including extubation would ensure timely patient care without compromising HCW safety and with minimal risk of facility contamination. Several improvised passive intubation shields or boxes have been reported, with significant limitations that make them likely ineffective and potentially harmful.[6][9-12] The research proposed in this application builds on our original device design that has addressed the shortcomings of aerosol boxes. This study will provide much needed knowledge about safe clinical use to build on the research team's simulation trials (research funded by the IWK Research Foundation Project Grant).

The device is designed to: (1) be simple and intuitive to use (2) be portable and rapidly deployed (3) provide ergonomic operator access (4) contain the spread of aerosols (5) permanently trap contaminants while minimizing the risk of aerosol resuspension during removal and room cleaning (6) be easily and safely disposed of and (7) inexpensive. Previous testing of the ease of use, potential safety implications and the impact on facility contamination has provided evidence that informs clinical evaluation in this study. Study findings may extend to health system management, public health response, decision-making and planning within and across jurisdictions in Canada and internationally.

This equivalence trial will aim to determine whether intubation with the flexible, disposable, active aerosol containment device is similar to intubation without the enclosure device with respect to intubation times, secondary safety endpoint and exploratory endpoints representing patient and anesthesiologist experiences and perceptions.

Objectives

The trial objective is to test ease of use in the operating room environment and patient safety (as indicated by the time to airway placement and change in oxygen saturation) of prototype (model versions 2 and 3, see description below) of an airborne pathogen containment device intended to decrease viral contamination during airway management. The testing will address the following research questions centered on the effect of physical presence of the device during the intubation process:

Q1: What is the difference in time to placement of airway (ta) with and without the containment device? Q2: Is the change in physiologic parameters upon airway placement significantly different in the presence of the device? [13][14] Q3: Does the use of the device affect the first attempt airway placement success rate? Q4: What is the impact on patients' and anesthesiologists' experience and satisfaction?

Trial endpoints Primary endpoint: Intubation times The null hypothesis states that intubation times with (experimental group) and without the containment device (standard treatment) differ by more than the equivalence margin of 10% (see sample size calculation).

Secondary endpoint: the number of patients experiencing either of the 2 co-secondary endpoints.

Co-secondary endpoint 1: Number of patients with post-intubation SaO2 <90% Co-secondary endpoint 2: The number of intubations requiring more than one attempt The 2 endpoints are not independent: requiring additional intubation attempts may lead to low SaO2 and positive pressure ventilation to maintain SaO2. Conversely, unduly persisting in 1st attempt may lead to low SaO2. These endpoints are thus complementary in capturing the potential effect of containment device. The benefit of combining them is avoidance of inflating the Type II error rate in controlling false discovery rate (which would be necessary with multiple endpoints).

The null hypothesis is that the number of patients with significant desaturation and/or multiple attempts will differ by more than the equivalence margin (see sample size calculation).

Exploratory endpoint 1: Absolute pre-post intubation change in end-tidal oxygen (change in ETCO2) Exploratory endpoint 2: Mean patient visual analogue scale (VAS) satisfaction score with the experience of "going to sleep" Exploratory endpoint 3: Mean anesthesiologist VAS "ease of airway management score"

Declaring device "success" or "failure" The trial can declare equivalence ("success") if statistical evidence is found to reject the null hypothesis for the primary endpoint of > 10% difference (equivalence margin) in intubation times.

It is, however, possible that the device does not meet the primary endpoint (the difference between intubation times is greater than the prespecified equivalence margin), but that the overall intubation times (at least 90% of the intubations) with device in place are within 60 seconds - a generally accepted "safe" intubation time. In this event, the device can still be deemed successful provided it meets the secondary (safety) endpoint. The secondary endpoint combines indicators that reflect adverse consequences of prolonged intubation time.

In the event that neither the primary nor the secondary endpoints are met, the device will have "failed" the clinical trial. The acquired data including exploratory endpoints and survey data will be reviewed and used to identify problems and, if possible, address them through device re-design.

ELIGIBILITY:
Inclusion Criteria:

* ASA class 1 and 2
* Elective surgery
* Adults >18 years of age
* Ability to give informed consent
* Surgery in supine or lithotomy position
* Surgical site: abdominal, pelvic, lower limb or distal upper limb
* Endotracheal intubation is indicated as per attending anesthesiologist

Exclusion Criteria:

* BMI >40
* pregnancy
* "full stomach" or increased intraabdominal pressure (as per attending anesthesiologist)
* predictors of difficult airway management as per attending anesthesiologist
* airway management plan (as per attending anesthesiologist) that is incompatible with study protocol
* initial ventilatory settings that are incompatible with planned care as per study protocol
* anxiety disorder (including claustrophobia)
* significant cardiovascular or respiratory disease (including pleural effusion, pulmonary edema, etc.)
* anticipated significant level of post-operative sedation preventing survey participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Duration of time needed to place an airway. | Day of surgery (intubation)
  Difference in means of airway times with and without the device present.

SECONDARY OUTCOMES:
Mean delta ETCO2 | For 5 min pre- and post- intubation
  End-tidal carbon dioxide (ETCO2) is the level of carbon dioxide that is released at the end of an exhaled breath.
First pass intubation success rate (%) | Day of Surgery - intubation
  Intubation - insertion of an endotracheal tube in a patient
Patient Body Mass Index | Day of Surgery
Blood Pressure | Every 1 minute during surgery (at least 2 measures taken prior to device deployment and 2 prior to induction)
  Systolic and diastolic blood pressure
Mean nadir ETO2 (%) | For 5 min pre- and post- intubation
  End-tidal Oxygen (ETO2) is the level of oxygen in the functional reserve capacity of the lungs.
Age | Day of surgery
  Age of the patient
Sex | Day of surgery
Incidence of SaO2 <90% | During time spent in surgical recovery room
  SaO2 is the percentage of oxygen-containing hemoglobin in the blood.
Time interval of laryngoscopy starting to 1st breath by endotracheal tube | Day of Surgery
  Laryngoscopy is a medical procedure where a doctor examines the back of the throat, voice box (larynx), and vocal cords using a special instrument called a laryngoscope.
Time interval of the patient leaving the operating room to being administered the patient feedback survey | Day of surgery
Time to achieving respiratory criteria for discharge from recovery room | Duration within the recovery room.
Patient feedback - Survey A | Administered within 24-hours of surgery
  The survey will seek input regarding patients' recollection of anxiety, comfort and overall acceptability prior to anesthesia induction and on emergence. Both cases and controls will be asked to answer the same questions. The aim of this part of the survey is to assess to what extent the presence of the device impacts patients' anesthesia experience. Part A questions were developed using a VAS for anxiety that has been validated in patients recovering from anesthesia. In addition, we will ask them to what extent they felt the team attended to their comfort and the overall satisfaction with their experience of the time period prior to anesthetic induction.
Patient Feedback - Survey B | Administered within 24-hours of surgery
  To answer device specific questions, patients in the control group will be shown a video of device deployment, placement on mannequin and disposal.
  In survey B, questions will be asked about perceived device benefits (patient safety, HCW safety) and downsides of adoption into anesthesia practice. The survey design will address domains outlined in the acceptability framework, but from the patients' perspectives. Part B questions have been used in the previous simulation trial's patient engagement survey. They had been developed through responses from testers who had viewed a similar video of the device in use. Both groups of patients will be asked to address the same aspects of device design and utility.
Years of experience of anesthesia provider | Day of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- IWK Health Centre, Halifax, Nova Scotia, Canada

REFERENCES:
- [Background] Fong S, Li E, Violato E, Reid A, Gu Y. Impact of aerosol box on intubation during COVID-19: a simulation study of normal and difficult airways. Can J Anaesth. 2021 Apr;68(4):496-504. doi: 10.1007/s12630-020-01825-y. Epub 2020 Oct 9. PMID 33033956
- [Background] Begley JL, Lavery KE, Nickson CP, Brewster DJ. The aerosol box for intubation in coronavirus disease 2019 patients: an in-situ simulation crossover study. Anaesthesia. 2020 Aug;75(8):1014-1021. doi: 10.1111/anae.15115. Epub 2020 Jun 1. PMID 32397008
- [Background] Labaste F, Ferre F, Combelles H, Rey V, Foissac JC, Senechal A, Conil JM, Minville V. Validation of a visual analogue scale for the evaluation of the postoperative anxiety: A prospective observational study. Nurs Open. 2019 Jul 11;6(4):1323-1330. doi: 10.1002/nop2.330. eCollection 2019 Oct. PMID 31660159
- [Background] Casey JD, Semler MW. Beginning of the End? End-tidal Oxygen as an Outcome in Airway Management Research. EClinicalMedicine. 2019 Jul 24;13:10-11. doi: 10.1016/j.eclinm.2019.07.006. eCollection 2019 Aug. No abstract available. PMID 31517257
- [Background] Wang J, Du G. COVID-19 may transmit through aerosol. Ir J Med Sci. 2020 Nov;189(4):1143-1144. doi: 10.1007/s11845-020-02218-2. Epub 2020 Mar 24. No abstract available. PMID 32212099
- [Background] Simpson JP, Wong DN, Verco L, Carter R, Dzidowski M, Chan PY. Measurement of airborne particle exposure during simulated tracheal intubation using various proposed aerosol containment devices during the COVID-19 pandemic. Anaesthesia. 2020 Dec;75(12):1587-1595. doi: 10.1111/anae.15188. Epub 2020 Jul 9. PMID 32559315